CLINICAL TRIAL: NCT04246788
Title: Intensive Robotic Rehabilitation in Children With Hemiparesia Using GEOSYSTEM
Acronym: RIPHIGEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2019 SARRET; 2019-A02218-49 (Other: 2019-A02218-49)
Record Dates: First submitted 2020-01-24; First posted 2020-01-29 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-04

CONDITIONS: Infantile Hemiplegia
Keywords: Infantile hemiplegia; Cerebral palsy; Intensive robotic rehabilitation
MeSH Terms: conditions — Hemiplegia; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 : experimental group (Experimental): 5 sessions per week of 30 minutes of robot-assisted rehabilitation with the G-EO system during two weeks
  Interventions: Other: Intensive robotic rehabilitation
- Cohort 2 : controle group (Active Comparator): 3 sessions per week of 30 minutes of classical physiotherapy during two weeks
  Interventions: Other: classical physiotherapy

INTERVENTIONS:
Other: Intensive robotic rehabilitation — 5 sessions per week of 30 minutes of robot-assisted rehabilitation with the G-EO system during two weeks
  Arms: Cohort 1 : experimental group
Other: classical physiotherapy — 3 sessions per week of 30 minutes of classical physiotherapy during two weeks
  Arms: Cohort 2 : controle group

SUMMARY:
Cerebral palsy is the most frequent motor deficiency in children. Among other, it can leads to spastic diplegia or hemiplegia. Walking abilities is an important skill to the families' point of view in term of independence in curent life. Improving the walking parameters has been the main objective in several studies of rehabilitation. The G-EO system is a last generation robot assisting gait training that can adjust cadence, walk lengh, ankle and hip angles and other walking parameters to movement captation. Its superiority in terms of walking abilities has been demonstrated in adults with stroke sequelae. Only one study was realized in pediatric patients with spastic diplegia with promising results. The investigators hypothesize that intensive robot-assited gait training using the G-EO system in hemiplegic children can improve their walking abilities.

DETAILED DESCRIPTION:
Objective :

Primary objective: To evaluate walking velocity with the GRAIL (gait real-time analysis and interactive lab) after intensive robot-assisted gait training using the G-EO system in hemiplegic children.

Secondary objectives :Other parameters that will be evaluate include:

* Endurance on the 6 minute walking test
* Joint angles and muscular contraction on the GRAIL
* Number of steps and travelled distance /24h, cardiac frequency and quality of sleep using actimeter bracelet
* Motor functions using the GMFM (Gross Motor Function Measure)
* Spasticity using the modified Ashworth scale
* The functional independence using the Functional Independence Measure (FIM™) for children,
* The quality of life using the Patient Global Impression (PGI-I)
* Muscular strength using the muscular testing cotation scale
* The musculo-squeletal and adipose composition using the peripherical quantitative computed tomography (pQCT)
* The cerebral area activation using functional MRI Study Type: Controlled randomized pilote study Number of centres: Monocentric study, University hospital of Clermont-Ferrand

Study procedure:

* Experimental group: 5 sessions per week of 30 minutes of robot-assisted rehabilitation with the G-EO system during two weeks
* Control group : 3 sessions per week of 30 minutes of classical physiotherapy during two weeks

Study evaluation:

T0 : before rehabilitation :

* Actimeter for 24h
* 6 min walking test
* GRAIL
* Modified Ashworth scale
* FIM for children
* GMFM
* Muscular testing scale
* pQCT
* fMRI

T1 : one month after rehabilitation :

* idem T0
* PGI-I questionnary Principal judgement criteria: Walking velocity Secondary judgement criteria: endurance, joint angles, number of steps and travelled distance per 24h, quality of sleep, cardiac frequency, spasticity, functional independence, motor functions, muscular strength, musculo-squeletal and adipose composition, brain activated areas.

Number of subjects:

* 20 patients in the experimental group
* 20 patients in the control group All patients enrolled in the control group will benefit of the GEOsystem rehabilitation at the end of the protocole

Inclusion criteria:

Hemiplegic children aged from 4 to 18 years, with a GMFCS (Gross Motor Function Classification System) score between I and III with lower limb involvement. Children must walk alone with or without aid at least 10 meters, must have acquired sitting position, must be able to understand simple orders to follow the rehabilitation program.

Non inclusion criteria:

No lower limb involvement, spasticity = 4 on the modified Ashworth scale, severe cardiorespiratory disease forbidding the rehabilitation program, orthopedic surgery or botulinic toxin injections in the last 6 months before the beginning of the study.

Study calendar:

* Starting inclusions: March 2020
* Experimental procedure: March 2020 to March 2021
* Data analyses and synthesis: April 2021 to Dember 2021

Statistical analyses Statistical analysis will be performed using Stata 13 software (Stata-Corp, College Station, TX) by an experimented statistician (Bruno Pereira) working in the university hospital of Clermont-Ferrand. A type-I error set at α=0.05 will be considered. Monovariate and multivariate analyses considering age as a covariable will be performed.

Ethical considerations This study has already been presented at the local ethical committee and will be presented in July 2019 at the national " comité de protection des personnes ". Written informed consent from both parents will be collected at the inclusion. This study will be in agreement with the declaration of Helsinki and the current regulations of clinical trials. It will be declared on the internet site "clinicaltrials.gov".

Expected results :

Intensive robot-assisted gait training using the G-EO system may improve the walking abilities in children with infantile hemiplegia and consequently improve their independence and quality of life. Musculo-squeletal parameters and profile of cerebral activated areas involved in praxia may also be modified by this intensive rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic children aged from 4 to 18 years
* GMFCS (Gross Motor Function Classification System) score between I and III with lower limb involvement.
* Children must walk alone with or without aid at least 10 meters, must have acquired sitting position, must be able to understand simple orders to follow the rehabilitation program.
* Free and informed consent of holders of parental authority and of the patient
* Affiliated to the social security system

Exclusion Criteria:

* No lower limb involvement,
* spasticity = 4 on the modified Ashworth scale,
* severe cardiorespiratory disease forbidding the rehabilitation program,
* orthopedic surgery or botulinic toxin injections in the last 6 months before the beginning of the study.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Gait speed | day 1
  gait speed assessed during a gait assessment session using the GRAIL system
Gait speed | day 21
  gait speed assessed during a gait assessment session using the GRAIL system
Gait speed | day 51
  gait speed assessed during a gait assessment session using the GRAIL system

SECONDARY OUTCOMES:
6 min. walk test (6-WT) | day 1
  endurance evaluation by 6 min. walk test (6-WT)
6 min. walk test (6-WT) | day 21
  endurance evaluation by 6 min. walk test (6-WT)
6 min. walk test (6-WT) | day 51
  endurance evaluation by 6 min. walk test (6-WT)
joint angles | day 1
  Joint amplitudes measured during gait assessment with the GRAIL
joint angles | day 21
  Joint amplitudes measured during gait assessment with the GRAIL
joint angles | day 51
  Joint amplitudes measured during gait assessment with the GRAIL
number of steps per 24h | day 1
  Number of steps per 24h, measured using a wristband actimeter which will be given to each child for 24 hours
number of steps per 24h | day 21
  Number of steps per 24h, measured using a wristband actimeter which will be given to each child for 24 hours
number of steps per 24h | day 51
  Number of steps per 24h, measured using a wristband actimeter which will be given to each child for 24 hours
travelled distance | day 1
  distance traveled per 24 hours, per 24h, measured using a wristband actimeter which will be given to each child for 24 hours
travelled distance | day 21
  distance traveled per 24 hours, per 24h, measured using a wristband actimeter which will be given to each child for 24 hours
travelled distance | day 51
  distance traveled per 24 hours, per 24h, measured using a wristband actimeter which will be given to each child for 24 hours
quality of sleep: wristband actimeter | day 1
  quality of sleep per 24 hours, per 24h, measured using a wristband actimeter which will be given to each child for 24 hours
quality of sleep: wristband actimeter | day 21
  quality of sleep per 24 hours, per 24h, measured using a wristband actimeter which will be given to each child for 24 hours
quality of sleep: wristband actimeter | day 51
  quality of sleep per 24 hours, per 24h, measured using a wristband actimeter which will be given to each child for 24 hours
cardiac frequency | day 1
  heart rate per 24 hours, per 24h, measured using a wristband actimeter which will be given to each child for 24 hours
cardiac frequency | day 21
  heart rate per 24 hours, per 24h, measured using a wristband actimeter which will be given to each child for 24 hours
cardiac frequency | day 51
  heart rate per 24 hours, per 24h, measured using a wristband actimeter which will be given to each child for 24 hours
Evaluation of spasticity | day 1
  Evaluation of spasticity by the modified Ashworth scale
Evaluation of spasticity | day 21
  Evaluation of spasticity by the modified Ashworth scale
Evaluation of spasticity | day 51
  Evaluation of spasticity by the modified Ashworth scale
functional independence | day 1
  Overall functional independence assessed with the MIF-Môme autonomy scale
functional independence | day 21
  Overall functional independence assessed with the MIF-Môme autonomy scale
functional independence | day 51
  Overall functional independence assessed with the MIF-Môme autonomy scale
motor functions | day 1
  Overall motor function evaluated with the EMFG
motor functions | day 21
  Overall motor function evaluated with the EMFG
motor functions | day 51
  Overall motor function evaluated with the EMFG
muscular strength | day 1
  Muscle strength will be measured with a quotation scale (1 to 5) for manual muscle testing
muscular strength | day 21
  Muscle strength will be measured with a quotation scale (1 to 5) for manual muscle testing
muscular strength | day 51
  Muscle strength will be measured with a quotation scale (1 to 5) for manual muscle testing
Body composition measurements | day 21
  fat body mass
Body composition measurements | day 51
  fat body mass
Body composition measurements | day 21
  lean body mass
Body composition measurements | day 51
  lean body mass
brain activated areas | day 21
  Functional brain connectivity analyzes by functional brain MRI
brain activated areas | day 51
  Functional brain connectivity analyzes by functional brain MRI

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Sarret, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont Ferrand, Clermont-Ferrand, Auvergne, France